CLINICAL TRIAL: NCT03451591
Title: LACunar Intervention (LACI-2) Trial-2: Assessment of Safety and Efficacy of Cilostazol and Isosorbide Mononitrate to Prevent Recurrent Lacunar Stroke and Progression of Cerebral Small Vessel Disease.
Brief Title: LACunar Intervention (LACI-2) Trial-2
Acronym: LACI-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: V6 06Feb2020; CS/15/5/31475 (Other Grant/Funding Number: British Heart Foundation); 2016-002277-35 (EudraCT Number); 14911850 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2017-11-14; First posted 2018-03-02 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Small Vessel Diseases; Stroke, Lacunar
Keywords: Cerebral Small Vessel Diseases; Stroke, Lacunar; Dementia; Alzheimer's disease
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Stroke, Lacunar; Dementia; Alzheimer Disease | interventions — Cilostazol

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to start one of four treatments; isosorbide mononitrate only; cilostazol only; both isosorbide mononitrate and cilostazol or neither isosorbide mononitrate nor cilostazol.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Isosorbide Mononitrate XL (ISMN) (Active Comparator): Oral Isotard® 25mg XL (Isosorbide Mononitrate) tablets. Oral Isotard® 25mg XL: Day 1-5 / 25mg daily morning dose. Day 6 to week 52 / 50mg daily morning dose. Week 53 / 25mg daily morning dose. Week 54 / NIL dose. Or Oral Isosorbide mononitrate (ISMN) non-XL 20mg tablets: Day 1-5 / 20mg daily evening dose. Day 6 to week 52 / 20mg twice daily morning & evening. Week 53 / 20mg daily morning dose. Week 54 / NIL dose.
  Interventions: Drug: Isosorbide Mononitrate XL (ISMN)
- Cilostazol (Active Comparator): Oral Cilostazol 100mg tablets. Day 1-5 / 50mg daily evening dose. Day 6-10 / 50mg twice daily morning & evening. Day 11-15 / 50mg daily morning dose & 100mg daily evening dose. Day 16 to week 52 / 100mg twice daily morning & evening. Week 53 / 50mg twice daily morning & evening. Week 54 / NIL dose.
  Interventions: Drug: Cilostazol
- ISMN XL and Cilostazol (Active Comparator): Oral Isotard® 25 mg XL (ISMN) and oral Cilostazol 100mg tablets. Day 1-5 / ISMN - 25mg daily evening dose / Cilostazol - NIL. Day 6-10 / ISMN - 50mg daily morning dose and Cilostazol - NIL. Day 11-15 / ISMN - 50mg daily morning dose / Cilostazol - 50mg daily evening dose. Day 16-20 / ISMN - 50mg daily morning dose and Cilostazol - 50mg twice daily morning & evening. Day 21-25 / ISMN - 50mg daily morning dose and Cilostazol - twice daily, 50mg morning & 100mg evening dose. Day 26-30 ISMN - 50mg daily morning dose and Cilostazol 100mg - twice daily morning & evening. Day 30 to week 52 / ISMN 50mg morning dose and Cilostazol 100mg - twice daily morning & evening. Week 53 / ISMN 25mg daily morning dose and Cilostazol 50mg twice daily morning & evening. Week 54 / NIL dose
  Interventions: Drug: ISMN XL and Cilostazol
- Neither ISMN nor cilostazol (Placebo Comparator): Neither isosorbide mononitrate nor Cilostazol is administered for the entire duration of the study.
  Interventions: Other: Neither ISMN nor cilostazol

INTERVENTIONS:
Drug: Isosorbide Mononitrate XL (ISMN) — Isosorbide mononitrate (ISMN), is an NO donating organic nitrate that enhances vasodilation, is widely used in ischaemic heart disease, and has no antiplatelet activity.
  Other Names: Isosorbide mononitrate non-XL (ISMN)
  Arms: Isosorbide Mononitrate XL (ISMN)
Drug: Cilostazol — Cilostazol is a phosphodiesterase 3-inhibitor (PDE3-inhibitor) that enhances the PGI2-cAMP system. It has weak antiplatelet effects (so low bleeding risk), reduces infarct size and reduces ageing-related decline in myelin repair in experimental models.
  Arms: Cilostazol
Drug: ISMN XL and Cilostazol — Cilostazol is a phosphodiesterase 3-inhibitor (PDE3-inhibitor) that enhances the PGI2-cAMP system. It has weak antiplatelet effects (so low bleeding risk), reduces infarct size and reduces ageing-related decline in myelin repair in experimental models. Isosorbide mononitrate (ISMN), is an NO donating organic nitrate that enhances vasodilation, is widely used in ischaemic heart disease, and has no antiplatelet activity.
  Other Names: isosorbide mononitrate non-XL and cilostazol
  Arms: ISMN XL and Cilostazol
Other: Neither ISMN nor cilostazol — Neither isosorbide mononitrate nor Cilostazol administered for the entire duration of the study.
  Arms: Neither ISMN nor cilostazol

SUMMARY:
About 35,000 people each year in the UK have a type of stroke, called 'lacunar' or 'small vessel' stroke, which is different to other common types of stroke and for which there is no proven treatment. It is thought that small vessel stroke is caused by damage to the lining of the tiny blood vessels deep inside the brain that stops them functioning normally. This not only causes stroke but, perhaps more importantly, causes problems with thinking and walking, possibly causing up to 45% of all dementias either on its own, or mixed with Alzheimer's disease (about 350,000 patients in the UK). Some drugs that are commonly used in other blood vessel diseases may help improve small vessel function and prevent worsening of brain damage. One drug (cilostazol) has been tested in patients with stroke in the Asia Pacific countries but not on dementia; the other drug (isosorbide mononitrate) is widely used in the UK for heart disease but not stroke. The investigators want to set up a clinical trial to test if the study methods are practical so that patients and trial centres can follow the procedures, and to confirm how many patients have more stroke-like symptoms or experience worsening of their thinking skills. This information is needed to be sure that a very large clinical trial to find out if these drugs can prevent worsening of small vessel disease will be possible.

DETAILED DESCRIPTION:
A quarter of all ischaemic strokes (about 35000 per annum in the UK) are lacunar (small vessel) in type, mainly caused by an intrinsic, non-atheromatous, non-cardioembolic disease of the small deep perforating cerebral arterioles. More diffuse cerebral small vessel disease also causes up to 45% of dementias (350,000+ patients estimated currently in the UK), either alone or in association with Alzheimer's disease. There is no proven treatment for cerebral small vessel disease: conventional antiplatelet drugs may be ineffective or even hazardous, whilst antihypertensive treatment and statins may not have an effect. The disease mechanism is poorly understood but endothelial dysfunction, blood-brain barrier failure and vessel stiffness appear to contribute to the pathogenesis. Promising data available for licensed drugs with relevant modes of action, cilostazol (>6000 stroke patients in the Asia Pacific Region) and isosorbide mononitrate (ISMN, widely used in cardiac disease) support their testing in cerebral small vessel disease. This trial will be an Phase IIb preparatory to Phase III, randomised, partial factorial, open label, blinded end-point trial, testing cilostazol, ISMN, both, or neither, to assess the feasibility of recruitment, drug tolerability, trial procedures, safety and event rates in 400 patients recruited in UK stroke centres and followed-up to one year (primary endpoint). This trial is preparatory to a large, definitive, Phase III randomised controlled trial to prevent recurrent lacunar stroke and progressive small vessel disease-related physical and cognitive impairments after lacunar stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical lacunar stroke syndrome.
* Brain scanning* with MR including diffusion imaging wherever possible, and obtained soon after the presentation with stroke, shows either:

  * a recent, relevant (in time and location) acute lacunar infarct on diffusion MR imaging1,
  * or, if no visible acute lacunar infarct on diffusion MR imaging2 then there is no competing pathology as a cause for stroke (e.g. no acute cortical infarct, no acute intra-cerebral haemorrhage, no stroke mimic such as tumour, subdural haematoma);
  * or, if only a CT brain scan is available2 as in section 3 above, then there is a small relevant (in age and location) subcortical infarct, or if no infarct then there is no competing pathology as a cause for stroke (e.g. no acute cortical infarct, no acute intra-cerebral haemorrhage, no stroke mimic such as tumour, subdural haematoma).

    1. Note that if there is no acute lacunar infarct on MR diffusion imaging but there is a recent-appearing lacunar infarct on FLAIR, T2, or T1 (i.e. no cavitation or ex-vacuo effect; may be slightly swollen, ill-defined edges; or scan in the few weeks before the stroke does not show a lesion but there is an acute lacunar infarct on MR T2, FLAIR, T1 scanning after the stroke in an appropriate area of the brain for symptoms), then the T2, FLAIR, T1 lesion may be counted as the acute lacunar infarct in the absence of a diffusion lesion. Similarly, on CT2 a recent relevant small subcortical infarct would not show cavitation or shrinkage/ex vacuo effect.
    2. Note that about a third of patients with a clinically definite lacunar syndrome do not have a corresponding recent infarct visible on MRI but should still be classed as 'lacunar stroke' if no other explanation can be found for the symptoms. The presence of a recent cortical infarct on FLAIR, T2, T1, the recent timing being indicated by the characteristics above, would count as a competing pathology.

Note that the complete absence of any abnormality on MR or CT brain imaging (no acute subcortical infarct or pre-existing SVD such as white matter hyperintensities, lacunes, etc.) while occasionally seen in lacunar stroke is unusual and should question the diagnosis of lacunar ischaemic stroke.

* Age > 30 years
* Independent in activities of daily living (modified Rankin ≤2)
* Capacity to give consent themselves

Exclusion Criteria:

* Other significant active neurological illness present since suffering stroke (e.g. recurrent seizures, multiple sclerosis, brain tumour). Well-controlled epilepsy present prior to the stroke, a single seizure at onset of the stroke or provoked seizure is not an exclusion.
* Requiring assistance with activities of daily living (Modified Rankin ≥3)
* Has been diagnosed as having dementia on formal clinical assessment
* Active cardiac disease (atrial fibrillation, myocardial infarction in past 6 months, active angina, symptomatic cardiac failure)
* Diagnosis of hypotension, defined as sitting systolic blood pressure less than 100mmHg
* Definite indication for (i.e. already prescribed) either trial medication, or definite contraindication to a trial drug as per SPCs - lactose intolerance is a contraindication to ISMN preparations which contain lactose monohydrate - (indication for or contraindication to one of the trial drugs still allows randomisation to the other trial drug)
* Unable to swallow tablets
* Bleeding tendency (e.g. known platelets<100, active peptic ulcer, history of intracranial haemorrhage such as subdural haematoma, subarachnoid haemorrhage, intracerebral haemorrhage, but not asymptomatic haemorrhagic transformation of infarction or a few microbleeds, taking anticoagulant medication)
* Planned surgery during the trial period including carotid endarterectomy. Note prior and apparently successful carotid endarterectomy (or other surgery) is not an exclusion criterion and patients who would otherwise be eligible but require endarterectomy first may be randomised after recovery from successful endarterectomy.
* Other concurrent life threatening illness
* Unlikely to be available for follow-up (e.g. moving outside or visitor to the area)
* History of drug overdose or attempted suicide or significant active mental illness
* Pregnant or breastfeeding women, women of childbearing age not taking contraception. Acceptable contraception in women of childbearing age is a "highly effective" contraceptive measure as defined by the Clinical Trials Facilitation Group (http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf) and includes combined (oestrogen and progesterone containing) or progesterone-only contraception associated with inhibition of ovulation, or intrauterine device or bilateral tubal occlusion. Contraception must be continued for up to 30 days after the end of the IMP dosing schedule.
* Prohibited medications to either trial drug (see sections 4.5 of the appended SPCs and protocol section 6.6.3, plus no anticoagulant drugs); (prohibited medications to one of the trial drugs still allows randomisation to the other trial drug).
* Renal impairment (creatinine clearance <25 ml/min)
* Hepatic impairment
* Current enrolment in another Clinical Trial of Investigational Medicinal Product (CTIMP); still in extended follow-up beyond the CTIMP primary outcome and no longer taking that trial's IMP is not an exclusion to enrolment in LACI-2.
* Unable to tolerate MRI or contraindication to MRI (Claustrophobia, Pacemaker)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M Wardlaw, MB ChB, Study Director — University of Edinburgh
Locations (1):
- Royal Infirmary, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wardlaw JM, Woodhouse LJ, Mhlanga II, Oatey K, Heye AK, Bamford J, Cvoro V, Doubal FN, England T, Hassan A, Montgomery A, O'Brien JT, Roffe C, Sprigg N, Werring DJ, Bath PM; Lacunar Intervention Trial-2 (LACI-2) Investigator Group. Isosorbide Mononitrate and Cilostazol Treatment in Patients With Symptomatic Cerebral Small Vessel Disease: The Lacunar Intervention Trial-2 (LACI-2) Randomized Clinical Trial. JAMA Neurol. 2023 Jul 1;80(7):682-692. doi: 10.1001/jamaneurol.2023.1526. PMID 37222252
- [Derived] Kwan J, Hafdi M, Chiang LLW, Myint PK, Wong LS, Quinn TJ. Antithrombotic therapy to prevent cognitive decline in people with small vessel disease on neuroimaging but without dementia. Cochrane Database Syst Rev. 2022 Jul 14;7(7):CD012269. doi: 10.1002/14651858.CD012269.pub2. PMID 35833913

RESULTS

PARTICIPANT FLOW:
Period: Randomisation
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol | Neither ISMN Nor Cilostazol
Started | 90 | 91 | 91 | 91
Completed | 90 | 91 | 91 | 91
Not Completed | 0 | 0 | 0 | 0
Period: SAE Reporting - Exposure to IMP
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol | Neither ISMN Nor Cilostazol
Started | 181 (The study has a 2x2 partial factorial design. This allows testing of both drugs when given alone and together. Participants were allocated into one of four treatment groups. However, as some participants were in a group which received both treatments simultaneously then the subgroups reported for IMP exposure include a count of both participants from the single and the combined treatment groups as the total number exposed to that IMP) | 182 (The study has a 2x2 partial factorial design. This allows testing of both drugs when given alone and together. Participants were allocated into one of four treatment groups. However, as some participants were in a group which received both treatments simultaneously then the subgroups reported for IMP exposure include a count of both participants from the single and the combined treatment groups as the total number exposed to that IMP) | 91 | 91
Completed | 181 | 182 | 91 | 91
Not Completed | 0 | 0 | 0 | 0
Period: Randomisation to 12 Month Follow Up
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol | Neither ISMN Nor Cilostazol
Started | 90 (Participants were allocated into one of four treatment groups. However, as some participants were in a group which received both treatments simultaneously then the subgroups reported for IMP exposure include a count of both participants from the single and the combined treatment groups as the total number exposed to that IMP (Factorial Design).) | 91 (Participants were allocated into one of four treatment groups. However, as some participants were in a group which received both treatments simultaneously then the subgroups reported for IMP exposure include a count of both participants from the single and the combined treatment groups as the total number exposed to that IMP(Factorial Design).) | 91 | 91
Completed | 70 | 70 | 81 | 87
Not Completed | 20 | 21 | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol | Neither ISMN Nor Cilostazol | Total
Number analyzed (Participants) | 90 | 91 | 91 | 91 | 363
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [56 to 72] | 64 [57 to 73] | 63 [56 to 72] | 64 [57 to 74] | 64 [56 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 27 | 30 | 112
  Male | 63 | 63 | 64 | 61 | 251
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Stroke onset to randomisation, days [Mean (Standard Deviation); unit: days] | 223.8 (409.8) | 217.8 (456.7) | 263.9 (614.7) | 192.9 (270.3) | 224.6 (453.8)
Stroke onset to randomisation <=100 days [Count of Participants; unit: Participants] | 54 | 53 | 46 | 53 | 206
Highest education level - postgraduate [Count of Participants; unit: Participants] | 5 | 6 | 10 | 6 | 27
Highest education level - undergraduate [Count of Participants; unit: Participants] | 8 | 9 | 9 | 11 | 37
Highest education level - A Level or Equivalent [Count of Participants; unit: Participants] | 8 | 14 | 14 | 18 | 54
Highest education level - O-level/GCSE or equivalent [Count of Participants; unit: Participants] | 34 | 30 | 27 | 23 | 114
Highest education level - Secondary School [Count of Participants; unit: Participants] | 34 | 32 | 31 | 32 | 129
Highest education level - Primary School [Count of Participants; unit: Participants] | 1 | 0 | 0 | 1 | 2
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 145 (18.1) | 145.2 (20.6) | 145.1 (19.3) | 142.7 (20.1) | 144.5 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Phase III Trial
Description: Feasibility of Phase III trial, i.e. that eligible patients can be identified correctly, in sufficient numbers, enrolled and >95% retained in follow-up at one year, to achieve feasibility target sample size recruitment and randomisation of 400 patients in 24 months in the UK.
Time Frame: 36 months (24 Months Recruitment + 12 months Follow Up)
Population: Number of participants at 12 months who did not complete follow up - because they refused, were lost to follow up or withdrawn
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol | Neither ISMN Nor Cilostazol
Number analyzed (Participants) | 90 | 91 | 91 | 91
Participants | 20 | 21 | 10 | 4

2. Secondary Outcome: Trial Medication Tolerability Measured by Number of Participants With Adherence to Medication at Half Dose or More at 1 Year
Description: It is estimated that in this trial 75% of patients will be able to tolerate trial medication, in at least half dose, up to one year after randomisation (i.e. less than 25% will stop trial medication completely through inability to tolerate the drugs).
Time Frame: 12 months
Population: Adherence to medication at half dose or more at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol
Number analyzed (Participants) | 90 | 91 | 91
Participants | 59 | 48 | 45

3. Secondary Outcome: Incidence of Treatment Emergent Adverse Effects [Safety]
Description: Safety - symptoms of systemic or intracranial bleeding, recurrent cerebral and systemic vascular events, and vascular and non-vascular causes of death will be collected. It is estimated that in this trial the absolute risk of death, including fatal haemorrhage, will not differ significantly (ie fall outside the upper 95% CI) from 2% per year on trial drugs versus no trial drugs, when given in addition to guideline drugs; and will not increase bleeding or ischaemic SVD lesions significantly (at the p<0.01 level) on MRI.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol | Neither ISMN Nor Cilostazol
Number analyzed (Participants) | 90 | 91 | 91 | 91
Participants | 1 | 2 | 0 | 1

4. Secondary Outcome: Treatment Efficacy - Percentage of Participants Experiencing an Event (Stroke, TIA, Myocardial Ischaemia, Cognitive Impairment and Dementia)
Description: It is estimated that in this trial the combined rate of recurrent stroke, MI, death, cognitive impairment and dependency will be 40-50% at one year after enrolment in order to detect modest but clinically-important reductions in poor outcomes.
  The study has a 2x2 partial factorial design. This allows testing of both drugs when given alone and together. Participants were allocated into one of four treatment groups. However, as some participants were in a group which received both treatments simultaneously then the subgroups reported for IMP exposure include a count of both participants from the single and the combined treatment groups as the total number exposed to that IMP
Time Frame: 12 months
Population: Clinical, functional, QoL and global outcomes at 12 months- Stroke/TIA, MI, Cognitive impairment, Dependency, Death. Data are number (%)
Measure: Count of Participants; unit: Participants
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol | Neither ISMN Nor Cilostazol
Number analyzed (Participants) | 181 | 182 | 89 | 91
Participants | 80 | 84 | 36 | 55

ADVERSE EVENTS:
Time Frame: From randomisation to 12 months.
Description: Other [Not Including Serious] Adverse Events were not monitored/assessed. These are reported as 0 in the table below.
Arm/Group | Isosorbide Mononitrate XL (ISMN) | Cilostazol | ISMN XL and Cilostazol | Neither ISMN Nor Cilostazol
All-Cause Mortality (participants affected / at risk) | 1/181 | 1/182 | 0/91 | 1/91
Serious Adverse Events (participants affected / at risk) | 21/181 | 29/182 | 15/91 | 12/91
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isosorbide Mononitrate XL (ISMN) (N=181) | Cilostazol (N=182) | ISMN XL and Cilostazol (N=91) | Neither ISMN Nor Cilostazol (N=91)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 7 (7) | 8 (8) | 5 (5) | 1 (1)
Genitourinary (Renal and urinary disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Haematological (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metabolic/Endocrine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infection/sepsis (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Tumour/ malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Other (General disorders) | 5 (5) | 6 (6) | 3 (3) | 4 (4)
Cardiovascular (Cardiac disorders) | 5 (5) | 7 (7) | 4 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
The open label design may have facilitated bias, though there is no evidence for this. The follow-up co-ordinators were masked to allocated drug whilst recording outcome data. Recruitment and one year follow-up at sites in LACI2 was affected by the SARS-Cov-19 pandemic. Some patients were unable to return for MRI or in person assessments at sites (Trails, BP) or return postal follow-up forms. As a factorial trial, comparison of the combination of drugs versus no drugs was underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03451591/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03451591/SAP_001.pdf